CLINICAL TRIAL: NCT07168928
Title: School-Based Nutrition Education and School Dietitian Model in Primary School Students: A Randomised Controlled Trial
Brief Title: School-Based Nutrition Education in Primary Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çağlar Akçalı (Other)
Responsible Party: Sponsor-Investigator, Çağlar Akçalı, Assistant Professor, Department of Nutrition and Dietetics, Faculty of Health Sciences, Mardin Artuklu University, Mardin Artuklu University
Organization: Mardin Artuklu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-7
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Childhood Obesity; School-Aged Children; Nutrition Education
Keywords: School-based nutrition education; school-aged children; nutrition knowledge; school dietitian; anthropometric measurements
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: This study used a randomized, parallel assignment design. Fourth-grade primary school students were randomly allocated to either an intervention group or a control group. The intervention group received an eight-week classroom-based nutrition education program led by dietitians, while their parents participated in a four-week parent-focused education program. The control group continued with routine school activities without additional nutrition education during the study period. Data were collected at baseline, immediately after the intervention, and at a two-month follow-up for the intervention group.
Who Masked: Outcomes Assessor
Masking Description: The study was conducted as a single-blind trial. Participants and intervention providers were aware of group assignments; however, the researcher responsible for outcome assessments and data analysis was blinded to group allocation to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - School-Based Nutrition Education (Experimental): Students in this group participated in an eight-week, classroom-based nutrition education programme led by a school dietitian. The sessions were interactive and age-appropriate, focusing on healthy eating, food groups, meal planning, and the risks of processed foods. In addition, parents received a four-week educational programme on child nutrition and healthy dietary practices.
  Interventions: Behavioral: School-Based Nutrition Education Program
- Control Group - Routine School Activities (No Intervention): Students in this group continued with their routine school curriculum without receiving additional nutrition education during the intervention period. After the study was completed, control group students were provided access to the nutrition education materials.

INTERVENTIONS:
Behavioral: School-Based Nutrition Education Program — The intervention consisted of an eight-week, school-based nutrition education programme delivered to fourth-grade students by a school dietitian. Sessions were conducted once per week and included interactive lectures, games, and educational activities focusing on healthy eating, food groups, balanced meals, and the risks of processed food consumption. In addition, parents of students in the intervention group received a four-week educational programme on child nutrition, meal planning, and healthy lifestyle practices.
  Arms: Intervention Group - School-Based Nutrition Education

SUMMARY:
This study aims to evaluate the effects of a school-based nutrition education program and the implementation of a school dietitian model on primary school students in Mardin, Türkiye. A total of 67 fourth-grade students were randomized into intervention (n=32) and control (n=35) groups. The intervention group received an eight-week classroom-based nutrition education program, while their parents received four weeks of parent-focused education. Outcomes were measured using the Nutrition Knowledge Test, Nutrition Attitude Scale, Nutrition Behavior Scale, Child Physical Activity Questionnaire, and anthropometric assessments including weight, height, BMI, and waist circumference. The study seeks to determine whether dietitian-led school-based nutrition education can improve children's nutrition knowledge, attitudes, and behaviours, as well as influence anthropometric measures. Findings from this trial are expected to inform future strategies for integrating school dietitians and structured nutrition education into primary schools in Türkiye.

DETAILED DESCRIPTION:
Childhood obesity and malnutrition are urgent public health challenges in Türkiye, particularly in regions with limited access to structured health promotion programmes. Schools represent an appropriate setting for preventive strategies as they provide consistent opportunities for health education and behaviour reinforcement.

Study Design and Randomisation This study was designed as a single-centre, parallel-group, randomised controlled trial (RCT) conducted in a public primary school in Mardin, Türkiye. A total of 70 fourth-grade students were recruited and randomly allocated into intervention and control groups using a simple randomisation procedure performed by an independent researcher. Allocation was concealed until group assignments were finalised.

Intervention The intervention group participated in an eight-week school-based nutrition education programme, led by a registered dietitian, with one session delivered per week during school hours. Each session lasted approximately 40 minutes and included structured modules on food groups, balanced diet, healthy snacking, and the risks of processed foods. Interactive teaching methods such as educational games, puzzles, and visual aids were applied to increase engagement. In parallel, parents of the intervention group students attended a four-week supplementary programme delivered in evening sessions, covering home-based nutrition practices and strategies for supporting healthy child eating behaviours.

The control group continued routine school activities during the study period. To ensure equity, they were provided with an abridged version of the nutrition education materials after study completion.

Data Collection Procedures Measurements were performed at three time points: baseline (T0), immediately after the intervention (T1), and two months post-intervention (T2). Trained assessors, blinded to group allocation, collected data following standardised protocols.

Instruments used included:

* Nutrition Knowledge Test (NKT)
* Nutrition Attitude Scale (NAS)
* Nutrition Behaviour Scale (NBS)
* Child Physical Activity Questionnaire (CPAQ)

Anthropometric data (height, weight, waist circumference, and BMI) were measured using calibrated equipment under uniform conditions.

Outcomes and Analysis Primary outcomes included changes in nutrition knowledge, attitudes, and behaviours, as well as physical activity levels. Secondary outcomes focused on anthropometric indicators and dietary habits. Data were analysed using intention-to-treat principles. Continuous variables were evaluated with repeated measures ANOVA to detect changes across the three assessment points, while categorical variables were tested with chi-square statistics. A p-value <0.05 was considered statistically significant.

Ethical and Quality Considerations Ethical approval was obtained from the institutional review board, and written informed consent was secured from parents alongside child assent. Confidentiality was maintained by anonymising data, and all educational materials were standardised to ensure consistency in intervention delivery.

Significance By providing a structured description of the intervention design and evaluation process, this study aims to generate evidence for the effectiveness of integrating school dietitians into the Turkish primary education system. The results will inform national strategies targeting childhood obesity prevention and promote sustainable health policies.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as a fourth-grade student in the selected primary school in Mardin, Türkiye.
* Aged between 10 and 11 years.
* Able to participate in classroom-based activities and complete the study assessments.
* Obtained written informed consent from parents.

Exclusion Criteria:

* Students with physical or cognitive impairments that prevent participation in educational sessions or completion of questionnaires.
* Absence from school during the intervention period that would preclude participation in the majority of sessions.

Ages: 10 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Nutrition Knowledge Score | Baseline, immediately post-intervention (8 weeks), and 2-month follow-up.
  In order to evaluate the nutritional behaviours, knowledge level and attitudes of the students, questions prepared by making use of the literature and in parallel with the nutrition education given were used. In the evaluation, +1 point was given for each correct answer, 0 points for each incorrect answer, and the total score was reported. Higher scores obtained from the test indicate higher nutritional knowledge.
Nutrition Attitude Score | Baseline, immediately post-intervention (8 weeks), and 2-month follow-up.
  The scale consists of exercise, nutrition, smoking and stress control sub-dimensions. In this study, only the 'nutrition' sub-dimension was used. The overall internal consistency coefficient of the scale was reported as 0.79 and the internal consistency coefficient of the nutrition subscale was reported as 0.68. The nutrition sub-dimension assesses the child's attitude towards behaviours to reduce fat intake, increase healthy food consumption and diets that support heart health. Scale items are scored between 1 (strongly disagree) and 4 (strongly agree) and the total score ranges from 4 to 16. The high scores obtained reflect favourable nutritional attitudes.
Nutrition Behaviour Score | Baseline, immediately post-intervention (8 weeks), and 2-month follow-up.
  It was developed to determine children's food preferences. It consists of 14 items featuring images of healthy and unhealthy foods. On the scale, each unhealthy food choice is assigned -1 point, each healthy food choice is assigned +1 point, and the total score ranges from -14 to +14. High scores indicate healthy eating habits.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Baseline, immediately post-intervention (8 weeks), and 2-month follow-up.
  Change in BMI (kg/m²) calculated from measured height and weight of participants. This will assess the effect of the nutrition education programme on growth and weight status.
Waist Circumference | Baseline, immediately post-intervention (8 weeks), and 2-month follow-up.
  Change in waist circumference (cm) measured using a standard anthropometric tape at the midpoint between the lower rib and iliac crest. This will evaluate central adiposity changes following the intervention.
Physical Activity Score | Baseline, immediately post-intervention (8 weeks), and 2-month follow-up.
  The questionnaire was used to determine the physical activity levels of the students. The Cronbach's alpha coefficient as 0.86. CPAQ was developed to assess the physical activity levels of children aged 8-14 years. The form is filled in by the child. The form consists of 10 questions and the physical activity status of the child in the last seven days is questioned with the form. Except for the question questioning the disease status of the questionnaire, each item is evaluated as 5 points and an activity score between 1-5 is found. '1' indicates low physical activity and '5' indicates high physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Mardin Artuklu University, Mardin, Artuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and ethical considerations related to the small sample size, which may increase the risk of participant identification

REFERENCES:
- [Background] Erdim L, Ergun A, Kuguoglu S. Reliability and validity of the Turkish version of the Physical Activity Questionnaire for Older Children (PAQ-C). Turk J Med Sci. 2019 Feb 11;49(1):162-169. doi: 10.3906/sag-1806-212. PMID 30764593
- [Background] Kowalski KC, Crocker PRE, Faulkner RA. Validation of the physical activity questionnaire for older children. Pediatr Exerc Sci. 1997;9(2):174-186.
- [Background] Crocker PR, Bailey DA, Faulkner RA, Kowalski KC, McGrath R. Measuring general levels of physical activity: preliminary evidence for the Physical Activity Questionnaire for Older Children. Med Sci Sports Exerc. 1997 Oct;29(10):1344-9. doi: 10.1097/00005768-199710000-00011. PMID 9346166
- [Background] Edmundson E, Parcel GS, Perry CL, Feldman HA, Smyth M, Johnson CC, Layman A, Bachman K, Perkins T, Smith K, Stone E. The effects of the child and adolescent trial for cardiovascular health intervention on psychosocial determinants of cardiovascular disease risk behavior among third-grade students. Am J Health Promot. 1996 Jan-Feb;10(3):217-25. doi: 10.4278/0890-1171-10.3.217. PMID 10163302
- [Background] Haney MÖ, Bahar Z. Çocuk kalp sağlığını geliştirme tutum ölçeği'nin geçerlik ve güvenirliği. Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi. 2014;7(2):92-97.
- [Background] Arvidson CR. Children's Cardiovascular Health Promotion Attitude Scale: An Instrument Development. Texas Woman's University; 1990